CLINICAL TRIAL: NCT01849575
Title: Direct VIsualiZAtion of Asymptomatic Atherosclerotic Disease for Optimum Cardiovascular Prevention. A Population Based Pragmatic Randomised Controlled Trial Within Västerbotten Intervention Programme (VIP) and Ordinary Care.
Brief Title: Visualization of Asymptomatic Atherosclerotic Disease for Optimum Cardiovascular Prevention
Acronym: VIPVIZA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Västerbotten County Council, Sweden (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VIPVIZA version 20121204
Record Dates: First submitted 2013-05-03; First posted 2013-05-08 (Estimated); Results first posted 2020-05-07 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Cardiovascular Diseases
Keywords: Ultrasonography; Cardiovascular diseases; Prevention; Risk communication; Risk assessment; Behavioral change
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The cleaned structured data which is generated from the original data and does not contain personal numbers (identity data) and is stored on an encrypted E: drive on a computer that is exclusively used for VIPVIZA by the data manager. Access only by the data manager with password. The password is only known by the data manager. It is also kept in a sealed envelope in the save of the Medical Faculty.
  For each sub-project, data on selected variables in the structured data base is exported to a researcher by the data manager after approval from the VIPVIZA steering group. Thus, the participants' identity is masked for the outcome assessors since they have nu access neither to the original or the structured data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): The intervention: Giving communication about risk of cardiovascular disease in the form of written and graphical information about silent atheroscslerosis measured by carotid ultrasound examination as carotid intima-media thickness, highlighted as vascular age, and plaque formation, visualized as a traffic light (green - no plaque, red - plaque).The ultrasound results are given to the study person and his/her physician, in addition to information about conventional risk factors for cardiovascular disease
  Interventions: Behavioral: Intervention
- Control (No Intervention): The comaparator is that the study person and his/her physician do not get any information about carotid ultrasound results on silent atherosclerosis. They are only informed about results of measured conventional CVD risk factors

INTERVENTIONS:
Behavioral: Intervention — Information about carotid ultrasound results to the participant and his/her primary care physician in the form of atherosclerosis highlighted graphically in color against normal vascular age patterns and as plaque formation. General information about atherosclerosis as a dynamic modifiable process and recommendation to follow clinical guidelines for risk factor control. After 2-4 weeks a follow-up call by a research nurse, to give additional information and reassurance, if needed. Identical information to the study participant is sent by post after 6 months.
  CVD risk factors are managed according to clinical guidelines within primary health care during the entire study period.
  Other Names: Information about ultrasound results
  Arms: Intervention

SUMMARY:
The purpose of VIPVIZA is to assess the impact of pictorial information about asymptomatic atherosclerotic disease to both physician and patient, for improving physicians' adherence to prevention guidelines and patient perception and understanding of the cardiovascular disease (CVD) risk and consequent motivation for prevention. The intervention effect is assessed by differences between randomization groups in the primaryboutcome Framingham Risk Score (FRS) and the secondary outcomes the Systematic COronary Risk Evaluation (SCORE) as well as changes in these scores after one, three and six years. Secondary outcomes are also atherosclerotic disease progression, as assessed by repeated carotid ultrasound examination after three and six years, as well as the prevalence of acute events and mortality after 10 years . Social, psychological and cognitive determinants of behavioral change as well as the intervention impact on novel biomarkers will also be explored.

DETAILED DESCRIPTION:
Project description

The main objective of this project is to contribute to improved primary prevention of cardiovascular disease through the provision of a visual image and pictorial report of atherosclerosis while still asymptomatic. The image and report are seen and discussed by both physician and patient in order to improve guideline adherence and patient perception and understanding of the CVD risk and consequent motivation for prevention. The specific objectives include: 1. To assess the prevalence of asymptomatic atherosclerotic disease in men and women through identification of carotid plaques and measurement of carotid intima-media thickness (CIMT), and to relate plaques and CIMT to clinically estimated CVD risk factors and risk scores; 2. To explore the impact of pictorial representations of atherosclerosis on physicians´ adherence to prevention guidelines, and on individuals' quality of life, preventive measures, risk factor control and progress of atherosclerotic disease over the course of three and six years, as well as on premature CVD morbidity and mortality over the course of 5 and 10 years; 3. To evaluate how individuals' social, psychological, and cognitive characteristics relate to health behaviours, atherosclerosis and CVD risk at baseline and progression of any atherosclerosis; 4. To investigate biomarkers in relation to CIMT and plaques at baseline, changes in conventional CVD risk markers and lifestyle, and progression of atherosclerosis.

Survey of the field Primary prevention of CVD often fails due to poor adherence among practitioners and patients to evidence-based prevention guidelines on effective modification of risk factors by lifestyle change and pharmacological treatment. Contributory factors include poor communication about the CVD risk by the physician and inaccurate risk perception among patients. The risk message is usually communicated verbally or numerically, while potentially more effective visual tools are seldom used. For the clinical assessment of CVD risk the FRS and the European SCORE are most widely used. However, evidence that their use translates into reduced CVD morbidity and mortality is scarce. These risk scores focus on high-risk individuals, despite 60-70% of all CVD events occurring among individuals at low or intermediate risk for CVD. They might also be too abstract to lead to accurate risk perception and to motivate individuals to take preventive actions; information alone seldom results in rational behavior modification. VIPVIZA takes a different approach from current practice for the prevention of CVD. Instead of being based solely on indirect risk factors, this project evaluates the atherosclerotic disease itself while it still is subclinical, providing improved assessment, communication and perception of the CVD risk and hence greater motivation for prevention. This is achieved with ultrasonography of medium sized arteries with assessment of CIMT and existing atherosclerotic plaques.

Design, setting and study population:

The study is a pragmatic randomised open-label controlled trial with blinded evaluators (PROBE). VIPVIZA is integrated in and added to the ordinary Västerbotten Intervention Programme (VIP). Individuals with at least one clinical CVD risk factor were invited to the VIPVIZA trial when they participated in VIP (n=4177), resulting in inclusion of 3532 participants. Baseline visits with ultrasound examinations were carried out from April 29 2013 to June 7 2016. Participants were consecutively and randomly allocated to two groups (intervention and control group) using a computer-generated randomization list. The ultrasound examinations in VIPVIZA at baseline as well as after three and six years are performed at the hospitals in the three cities/towns (Umeå, Skellefteå, Lycksele), and in remote rural areas at primary health care centres. Risk factor measurements and questionnaires at follow-up after one, three and six years are carried out for participants living in Umeå at the Clinical Research Centre at Umeå University Hospital, and for participants in the rest of the county at their local primary health care center. Both groups are managed according to clinical guidelines for CVD prevention within primary care (not by the study team).

Intervention At baseline, pictorial representation of the carotid ultrasound results was given to each participant in the intervention group and their primary care physician. Atherosclerosis was presented as vascular age, with a gauge ranging from green through yellow, orange and red to illustrate the individual's biological age compared to chronological,age. A red or a green circle, like a traffic light, illustrated detected or no detected plaque, respectively. Brief written information about atherosclerosis as a dynamic process that is modifiable by a healthy lifestyle and pharmacological treatment, an interpretation of the result and general advice on CVD prevention were included. After 2-4 weeks, participants received a follow-up phone call by a research nurse in order to reassure and give additional information as needed. The same pictorial information was repeated to participants after 6 months. No information about the ultrasound result was given to the control group and their physicians.

At three- and six-year follow-up both the intervention and the control group participants and their respective primary care physician receive information about ultrasound results with the same format as was given to the intervention group at baseline. Thus, the intervention is completed at the time-point for three-year follow-up. After that the two groups are continuously followed through registries and compared with respect to atherosclerosis development and hard outcomes.

Data collection:

Clinical risk factors for cardiovascular disease: Measured at the baseline VIP health survey, at 1-, 3- and 6-year follow-up (blood pressure, lipids, and glucose, BMI and waist circumference).

Questionnaires: The VIP questionnaire covers health, socioeconomic situation, quality of life (RAND 36), lifestyle (physical activity, tobacco and alcohol consumption, diet), working conditions, social network. Validated psychometric instruments at baseline and 3-year follow-up included health literacy, coping strategies, an optimism-pessimism scale, self-efficacy, HADS and self-rated risk of CVD. Perceptions about preventive medication and a stress questionnaire at the 3-year follow-up. At 3-year follow-up questions on health literacy, coping strategies and optimism/pessimism are replaced by questionnaires on personality and dental care.

Carotid ultrasound examinations are performed at baseline, after 3 and6 years according to a standardized protocol.

Interviews: With subsamples of participants after the first, second and third ultrasound examination, and with primary care physicians after the first ultrasound examination.

Stored samples of blood to the Medical Biobank: This is done at the baseline VIP visit and at 3- and 6-year follow-up among participants, to be used for analyses of novel biomarkers Register data: Prescriptions, visits and risk factor measurements from the medical records system in Västerbotten County. Dental health and dental radiological examinations from Dental care. The Prescriptions register, Hospitalizations register and Causes of deaths register at the National Board of Health and Welfare. In addition, physical and psychological functioning and blood-group at military patterning at age around 18 from the Conscripts registry (for male participants only), educational level and income from Statistics Sweden and air pollutants by geographical region in the County of Västerbotten.

Time plan The study progress is largely according to the plan. Baseline examinations were conducted April 2013-June 2016, the 1-year follow-up examinations June 2014-August 2017, and the 3-year examinations September 2016 - June 2019. The six-year follow-up examinations started December 2019 which is a delay of 6 months due to administrative reasons. Register data from medical records, Statistics Sweden, the Conscripts register, Air-borne pollutants are underway April 2020. Data on morbidity and mortality will be retrieved in 2027, i.e. one year later than 10 years after trial start due to delay until data on events has been entered into the registries.

Ethical approval:

Study protocol version 4.0:

The VIPIVZA trial: Dnr 2011-445-32M date Feb 7 2012. Amendment 1: Dnr 2012-463-32M date December 19 2012. Amendment 2: Dnr 2013 373-32M date October 15 1013. Amendment 3: Dnr 2016-245-32M date May 31 2016. Amendment 4: Dnr 2017-95-32M date February 27 2017. Amendment 5: Dnr 2018-182-32 date May 28 2018.

Study protocol version 5.0:

Amendment 6: Dnr 2018-482-32M Date December 27 2018. Amendment 7: Dnr 2019-04619 Date September 24 2019.

ELIGIBILITY:
Inclusion Criteria:

- Participant in the Västerbotten Intervention Programme

and

* 40 years old and a history of CVD at age < 60 years among first-degree relative

or

* 50 years old and at least one of the following six criteria:
* a history of CVD at age < 60 years among first-degree relative,
* smoking,
* diabetes,
* hypertension,
* S-LDL-cholesterol ≥4.5 mmol/L,
* abdominal obesity

or

* 60 years old

Exclusion Criteria:

* Stenosis ≥50% of the carotid lumen

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3532 (Actual)
Dates: Start 2013-04-07 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2027-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Patrik Wennberg, MD, PhD, Principal Investigator — Umeå University; Ulf Näslund, Professor,MD, Principal Investigator — Umeå University Hospital
Locations (1):
- Clinical Reseach Center Umeå University Hospital, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vanoli D, Lindqvist P, Wiklund U, Henein M, Naslund U. Fully automated on-screen carotid intima-media thickness measurement: a screening tool for subclinical atherosclerosis. J Clin Ultrasound. 2013 Jul-Aug;41(6):333-9. doi: 10.1002/jcu.22041. Epub 2013 Mar 28. PMID 23553729
- [Result] Vanoli D, Wiklund U, Lindqvist P, Henein M, Naslund U. Successful novice's training in obtaining accurate assessment of carotid IMT using an automated ultrasound system. Eur Heart J Cardiovasc Imaging. 2014 Jun;15(6):637-42. doi: 10.1093/ehjci/jet254. Epub 2013 Dec 29. PMID 24378482
- [Result] Nyman E, Lindqvist P, Naslund U, Gronlund C. Risk Marker Variability in Subclinical Carotid Plaques Based on Ultrasound is Influenced by Cardiac Phase, Echogenicity and Size. Ultrasound Med Biol. 2018 Aug;44(8):1742-1750. doi: 10.1016/j.ultrasmedbio.2018.03.013. Epub 2018 May 4. PMID 29735317
- [Result] Naslund U, Ng N, Lundgren A, Fharm E, Gronlund C, Johansson H, Lindahl B, Lindahl B, Lindvall K, Nilsson SK, Nordin M, Nordin S, Nyman E, Rocklov J, Vanoli D, Weinehall L, Wennberg P, Wester P, Norberg M; VIPVIZA trial group. Visualization of asymptomatic atherosclerotic disease for optimum cardiovascular prevention (VIPVIZA): a pragmatic, open-label, randomised controlled trial. Lancet. 2019 Jan 12;393(10167):133-142. doi: 10.1016/S0140-6736(18)32818-6. Epub 2018 Dec 3. PMID 30522919
- [Result] Nyman E, Vanoli D, Naslund U, Gronlund C. Inter-sonographer reproducibility of carotid ultrasound plaque detection using Mannheim consensus in subclinical atherosclerosis. Clin Physiol Funct Imaging. 2020 Jan;40(1):46-51. doi: 10.1111/cpf.12602. Epub 2019 Oct 29. PMID 31605665
- [Result] Lindahl B, Norberg M, Johansson H, Lindvall K, Ng N, Nordin M, Nordin S, Naslund U, Persson A, Vanoli D, Schulz PJ. Health literacy is independently and inversely associated with carotid artery plaques and cardiovascular risk. Eur J Prev Cardiol. 2020 Jan;27(2):209-215. doi: 10.1177/2047487319882821. Epub 2019 Oct 15. PMID 31615294
- [Result] Bengtsson A, Lindvall K, Norberg M, Fharm E. Increased knowledge makes a difference! - general practitioners' experiences of pictorial information about subclinical atherosclerosis for primary prevention: an interview study from the VIPVIZA trial. Scand J Prim Health Care. 2021 Mar;39(1):77-84. doi: 10.1080/02813432.2021.1882083. Epub 2021 Feb 11. PMID 33569981
- [Result] Sjolander M, Carlberg B, Norberg M, Naslund U, Ng N. Prescription of Lipid-Lowering and Antihypertensive Drugs Following Pictorial Information About Subclinical Atherosclerosis: A Secondary Outcome of a Randomized Clinical Trial. JAMA Netw Open. 2021 Aug 2;4(8):e2121683. doi: 10.1001/jamanetworkopen.2021.21683. PMID 34410393
- [Result] Schulz PJ, Lindahl B, Hartung U, Naslund U, Norberg M, Nordin S. The right pick: Does a self-assessment measurement tool correctly identify health care consumers with inadequate health literacy? Patient Educ Couns. 2022 Apr;105(4):926-932. doi: 10.1016/j.pec.2021.07.045. Epub 2021 Jul 29. PMID 34366227
- [Result] Kovrov O, Landfors F, Saar-Kovrov V, Naslund U, Olivecrona G. Lipoprotein size is a main determinant for the rate of hydrolysis by exogenous LPL in human plasma. J Lipid Res. 2022 Jan;63(1):100144. doi: 10.1016/j.jlr.2021.100144. Epub 2021 Oct 26. PMID 34710432
- [Result] Holmberg H, Sjolander M, Glader EL, Naslund U, Carlberg B, Norberg M, Sjalander A. Time to initiation of lipid-lowering drugs for subclinical atherosclerosis: sub-study of VIPVIZA randomized controlled trial, with single-arm cross-over. Eur Heart J Open. 2022 Feb 4;2(1):oeac003. doi: 10.1093/ehjopen/oeac003. eCollection 2022 Jan. PMID 35919662
- [Result] Sommar JN, Norberg M, Gronlund C, Segersson D, Naslund U, Forsberg B. Long-term exposure to particulate air pollution and presence and progression of carotid artery plaques - A northern Sweden VIPVIZA cohort study. Environ Res. 2022 Aug;211:113061. doi: 10.1016/j.envres.2022.113061. Epub 2022 Mar 4. PMID 35257687
- [Result] Nyman E, Liv P, Wester P, Naslund U, Gronlund C. Carotid wall echogenicity at baseline associates with accelerated vascular aging in a middle-aged population. Int J Cardiovasc Imaging. 2023 Mar;39(3):575-583. doi: 10.1007/s10554-022-02760-3. Epub 2023 Jan 21. PMID 36680684
- [Result] Nyman E, Gronlund C, Vanoli D, Liv P, Norberg M, Bengtsson A, Wennberg P, Wester P, Naslund U; VIPVIZA trial group. Reduced progression of carotid intima media thickness by personalised pictorial presentation of subclinical atherosclerosis in VIPVIZA-A randomised controlled trial. Clin Physiol Funct Imaging. 2023 Jul;43(4):232-241. doi: 10.1111/cpf.12811. Epub 2023 Jan 27. PMID 36642849
- [Result] Andersson EM, Johansson H, Nordin S, Lindvall K. Cognitive and emotional reactions to pictorial-based risk communication on subclinical atherosclerosis: a qualitative study within the VIPVIZA trial. Scand J Prim Health Care. 2023 Mar;41(1):69-80. doi: 10.1080/02813432.2023.2178850. Epub 2023 Feb 28. PMID 36855328
- [Result] Naslund U, Norberg M, Wennberg P. The TANSNIP-PESA trial is not the end of the story. Eur Heart J. 2023 May 1;44(17):1574. doi: 10.1093/eurheartj/ehad135. No abstract available. PMID 36951199
- [Result] Fortuin-de Smidt M, Bergman F, Gronlund C, Hult A, Norberg M, Wennberg M, Wennberg P. Early adulthood exercise capacity, but not muscle strength, associates with subclinical atherosclerosis 40 years later in Swedish men. Eur J Prev Cardiol. 2023 Mar 27;30(5):407-415. doi: 10.1093/eurjpc/zwad007. PMID 36631734
- [Result] Ali H, Näslund U, Nyman E, Grönlund C. Translation of atherosclerotic disease features onto healthy carotid ultrasound images using domain-to-domain translation. Biomedical Signal Processing & Control. 2023
- [Result] Bengtsson A, Nyman E, Gronlund C, Wester P, Naslund U, Fharm E, Norberg M. Multi-view carotid ultrasound is stronger associated with cardiovascular risk factors than presence of plaque or single carotid intima media thickness measurements in subclinical atherosclerosis. Int J Cardiovasc Imaging. 2023 Aug;39(8):1461-1471. doi: 10.1007/s10554-023-02868-0. Epub 2023 May 30. PMID 37249653
- [Result] Nordin S, Norberg M, Braf I, Johansson H, Lindahl B, Lindvall K, Nordin M, Nyman E, Vallstrom C, Wennberg P, Liv P, Naslund U. Associations between emotional support and cardiovascular risk factors and subclinical atherosclerosis in middle-age. Psychol Health. 2025 Jun;40(6):997-1011. doi: 10.1080/08870446.2023.2286296. Epub 2023 Nov 23. PMID 37994844
- [Result] Salvador D Jr, Liv P, Norberg M, Pahud de Mortanges A, Saner H, Glisic M, Nicoll R, Muka T, Nyman E, Bano A, Naslund U. Changes in fasting plasma glucose and subclinical atherosclerosis: A cohort study from VIPVIZA trial. Atherosclerosis. 2024 Jul;394:117326. doi: 10.1016/j.atherosclerosis.2023.117326. Epub 2023 Oct 17. PMID 37932189
- [Derived] Sonnerstam E, Holmberg H, Carlberg B, Norberg M, Sjalander A, Glader EL. Beliefs about medicines in relation to the initiation of cardiovascular preventive medications during a 3 year follow-up period after inclusion in the VIPVIZA trial: a cohort study. BMJ Open. 2025 Dec 23;15(12):e100924. doi: 10.1136/bmjopen-2025-100924. PMID 41436264
- [Derived] Norberg M, Liv P, Naslund U, Wester P, Andersson EM, Nordin S. The Path for Men from Young Adulthood Results of Cognitive Tests to Subclinical Atherosclerosis at Age 60: The Mediating Role of Socioeconomic Status, Lifestyle and Cardiovascular Disease Risk Factors-Results from a VIPVIZA Study. Rev Cardiovasc Med. 2025 Mar 20;26(3):26312. doi: 10.31083/RCM26312. eCollection 2025 Mar. PMID 40160597
- [Derived] Soderstrom M, Gronlund C, Liv P, Nyman E, Naslund U, Wester P. Aortic arterial stiffness associates with carotid intima-media thickness and carotid plaques in younger middle-aged healthy people. Blood Press. 2024 Dec;33(1):2405161. doi: 10.1080/08037051.2024.2405161. Epub 2024 Sep 18. PMID 39291635
- [Derived] Holmberg H, Glader EL, Naslund U, Carlberg B, Sonnerstam E, Norberg M, Sjalander A. Improved adherence to statin treatment and differences in results between men and women after pictorial risk communication-a sub-study of the VIPVIZA RCT. Eur J Clin Pharmacol. 2024 Aug;80(8):1209-1218. doi: 10.1007/s00228-024-03694-6. Epub 2024 Apr 29. PMID 38684558
- [Derived] Andersson EM, Lindvall K, Wennberg P, Johansson H, Nordin S. From risk communication about asymptomatic atherosclerosis to cognitive and emotional reactions and lifestyle modification. BMC Psychol. 2024 Jan 24;12(1):47. doi: 10.1186/s40359-023-01467-x. PMID 38268015

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Information and collection informed consent: April 11 2012- June 1 2016 at the occasion of participation in the Västerbotten Intervention Program, Sweden, an ongoing CVD prevention program targeting residents at ages 40, 50 and 60 years
  Inclusion in the trial: April 29 2013-June 7 2016 at the Clinical research center, Umea University Hospital
Groups:
- Intervention: Intervention: Information about carotid ultrasound results to the participant and his/her primary care physician. Carotid intima-media thickness was presented as vascular age illustrating the individual's biological compared to chronological age, with a gauge going from green (at least 10 years younger), to yellow, orange or red (at least 10 years older). Plaque formation was a traffic light (green - no plaque, red - plaque). General information about atherosclerosis as a dynamic modifiable process and recommendation to follow clinical guidelines for risk factor control. After 2-4 weeks a follow-up call by a research nurse, to give additional information and reassurance, if needed. Identical information to the study participant is sent by post after 6 months.
  CVD risk factors are managed according to clinical guidelines within primary health care during the entire study period.
- Control: The comaparator is that the study person and his/her physician do not get any information about carotid ultrasound results on silent atherosclerosis. They are only informed about results of measured conventional CVD risk factors CVD risk factors are managed according to clinical guidelines within primary health care during the entire study period.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 1749 | 1783
Completed | 1599 | 1576
Not Completed | 150 | 207

BASELINE CHARACTERISTICS:
Groups:
- Intervention: Intervention: Pictorial information about carotid ultrasound results to the participant and his/her primary care physician. Asymptomatic atherosclerosis presented as vascular age with a gauge going from green (biological age 10 years younger than chronological age), over yellow, orange to red (10 years older). Plaque formation shown as a traffic light with a green dot (no plaque) or red dot (plaque) for each side. General information about atherosclerosis as a dynamic modifiable process and recommendation to follow clinical guidelines for risk factor control. After 2-4 weeks a follow-up call by a research nurse, to give additional information and reassurance, if needed. Identical information to the study participant is sent by post after 6 months.
  CVD risk factors are managed according to clinical guidelines within primary health care during the entire study period.
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 1749 | 1783 | 3532
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1749 | 1783 | 3532
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 940 | 930 | 1870
  Male | 809 | 853 | 1662
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Region Västerbotten, Sweden
  participants
    Sweden | 1749 | 1783 | 3532
Framingham Risk Score [Mean (Standard Deviation); unit: % risk of CVD within 10 years] — Composite gender-specific algorithm used to estimate the 10-year cardiovascular risk (%) of an individual, based on levels of blood pressure, total cholesterol, LDL-cholesterol, systolic blood pressure, treatment for high blood pressure, diabetes, smoking and age.
  This 10-year risk is evaluated as a continuous variable or categorized into five categories: Low risk (<5%), Light risk (5-9%), Moderate risk (10-19%), High risk (20-39%), Very high risk (>=40%)
  % risk of CVD within 10 years | 12.9 (9.6) | 12.8 (9.1) | 12.9 (9.3)

OUTCOME MEASURES:

1. Primary Outcome: FRS
Description: Framingham risk score. Composite gender-specific algorithm used to estimate the 10-year cardiovascular risk of an individual, based on levels of blood pressure, total cholesterol, LDL-cholesterol, systolic blood pressure, treatment for high blood pressure, diabetes, smoking and age. Minimum value=0, maximum value 100. Higher score means a worse outcome, i.e. a higher risk of cardiovascular diseases.
Time Frame: one year
Measure: Number (99.5% Confidence Interval); unit: % risk of a CVD event within 10 years
Groups:
- Intervention: The intervention: Giving communication about risk of cardiovascular disease in the form of written and graphical information about silent atheroscslerosis measured by carotid ultrasound examination as carotid intima-media thickness, highlighted as vascular age, and plaque formation, visualized as a traffic light (green - no plaque, red - plaque).The ultrasound results are given to the study person and his/her physician, in addition to information about conventional risk factors for cardiovascular disease
  Intervention: Information about carotid ultrasound results to the participant and his/her primary care physician in the form of atherosclerosis highlighted graphically in color against normal vascular age patterns and as plaque formation. General information about atherosclerosis as a dynamic modifiable process and recommendation to follow clinical guidelines for risk factor control. After 2-4 weeks a follow-up call by a research nurse, to give additional information and reassurance, if needed. Identical information to the study participant is sent by post after 6 months.
  CVD risk factors are managed according to clinical guidelines within primary health care during the entire study period.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1599 | 1576
% risk of a CVD event within 10 years | 12.2 [11.6 to 12.9] | 13.3 [12.6 to 14.0]

2. Secondary Outcome: SCORE
Description: SCORE: European systematic coronary risk evaluation. Risk of death (%) in myocardial infarction within 10 years expressed as statistical assessment based on smoking, systolic blood-pressure, blood cholesterol, age and sex.
  SCORE is evaluated as a continuous variable with Minimum value=0%, maximum value=100%. Higher score means a worse outcome, i.e. a higher risk of cardiovascular diseases.
Time Frame: Follow-up after one year
Measure: Number (99.5% Confidence Interval); unit: % risk of a CVD event within 10 years
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1749 | 1783
% risk of a CVD event within 10 years | 1.42 [1.33 to 1.55] | 1.58 [1.47 to 1.68]

3. Secondary Outcome: Hospitalizations Due to Stroke, Myocardial Infarctions and Re-vascularizations
Description: Data will be collected from the In-patient registry at the National Board of Health and Welfare.
Time Frame: 10 years
Reporting Status: Not Posted, anticipated posting 2027-12

4. Secondary Outcome: Total Mortality and Cause-specific Mortality Due to Myocardial Infarctions and Stroke
Description: Data will be collected from the Causes of Deaths registry at the National Board of Health and Welfare.
Time Frame: 10 years
Reporting Status: Not Posted, anticipated posting 2027-12

5. Secondary Outcome: Total Mortality
Description: Data will be collected from computerized medical records from hospital care in the county, regional quality registry on myocardial infarctions and from the In-patient registry at the National Board of Health and Welfare.
Time Frame: 10 years
Reporting Status: Not Posted, anticipated posting 2027-12

6. Secondary Outcome: Carotid Atherosclerosis
Description: Carotid intima media thickness
Time Frame: 3 years after baseline
Population: All participants who completed the carotid ultrasound examination at the 3-year follow-up
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1575 | 1579
mm | 0.680 (0.151) | 0.685 (0.165)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.001, ANCOVA

7. Other Pre Specified Outcome: FRS, Adjusted for Baseline Values
Description: FRS=Framingham risk score. Composite gender-specific algorithm used to estimate the 10-year cardiovascular risk of an individual, based on levels of blood pressure, total cholesterol, LDL-cholesterol, systolic blood pressure, treatment for high blood pressure, diabetes, smoking and age. Minimum value=0, maximum value 100. Higher score means a worse outcome, i.e. a higher risk of cardiovascular diseases.
Time Frame: Follow-up after three years during September 5 2016 - May 28 2019
Measure: Number (95% Confidence Interval); unit: % risk of a CVD event within 10 years
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1580 | 1587
% risk of a CVD event within 10 years | 13.33 [13.02 to 13.64] | 14.13 [13.83 to 14.44]

8. Other Pre Specified Outcome: SCORE Adjusted for Baseline Levels
Description: as for outcome 2
Time Frame: Three years of follow-up, data collected during September 5 2016 - May 28 2019
Measure: Number (95% Confidence Interval); unit: % risk of a CVD event within 10 years
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1580 | 1587
% risk of a CVD event within 10 years | 1.69 [1.64 to 1.74] | 1.83 [1.78 to 1.88]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 5/1749 | 2/1783
Serious Adverse Events (participants affected / at risk) | 0/1749 | 0/1783
Other Adverse Events (participants affected / at risk) | 50/1749 | 0/1783
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=1749) | Control (N=1783)
Anxiety (Psychiatric disorders) | 50 (50) | 0 (0) — Anxiety due to information about subclinical atherosclerosis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (5):
  • Study Protocol (2023-12-12): https://cdn.clinicaltrials.gov/large-docs/75/NCT01849575/Prot_009.pdf
  • Statistical Analysis Plan: Primary outcome from base line up to one year of follow up (2018-05-28): https://cdn.clinicaltrials.gov/large-docs/75/NCT01849575/SAP_004.pdf
  • Statistical Analysis Plan: Secondary outcomes up to 10 years of follow-up (2019-10-27): https://cdn.clinicaltrials.gov/large-docs/75/NCT01849575/SAP_007.pdf
  • Statistical Analysis Plan: Evaluation after 6 years (2024-01-12): https://cdn.clinicaltrials.gov/large-docs/75/NCT01849575/SAP_010.pdf
  • Informed Consent Form (2018-05-29): https://cdn.clinicaltrials.gov/large-docs/75/NCT01849575/ICF_006.pdf